CLINICAL TRIAL: NCT03891706
Title: An Open, Single-center, Stage I Clinical Study of Individualized Tumor Specific TCR-T Cells in the Treatment of Advanced Solid Tumors.
Brief Title: Individualized Tumor Specific TCR- T Cells in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou FineImmune Biotechnology Co., LTD. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FI-FIT001-001
Record Dates: First submitted 2019-03-24; First posted 2019-03-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: TCR-T
MeSH Terms: interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TCR-T cell infusion (Experimental): Patient will exposed to Individualized Tumor-t Cell Receptor (TCR) -Mediated T Cells therapy
  Interventions: Drug: tumor-specific TCR-T cells; Drug: Interleukin-2

INTERVENTIONS:
Drug: tumor-specific TCR-T cells — On day 0 and day 14, 0.5-5x10^9 TCR-T cells will be infused intravenously (IV) over 1 hour,patients may choose to receive more cell infusions if they benefit from the treatment.
  Other Names: TCR-T cells; FIT-001
Drug: Interleukin-2 — Aldesleukin 3,000,000 IU. IV.QD beginning within 24 hours of cell infusion and continuing for up to 5 days .
  Other Names: IL-2

SUMMARY:
The primary purpose of this study is to evaluate the safety of the tumor-specific TCR-T cells in the treatment of advanced Solid Tumor .

The secondary purpose of this study is to preliminarily showed the effect of TCR-T cells in the treatment of advanced Solid Tumor .

DETAILED DESCRIPTION:
This study is an open, single-center, phase I clinical trial which is aim to evaluate the safety and tolerability of tumor-specific TCR-T cells. In this study, these TCR-T cells will be multiplied, or grown, in the laboratory.Subjects will received TCR-T cells infusions twice at day 0 and day 14, with the use of IL-2 for 5 consecutive days after every cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old, regardless of gender;
2. Diagnosed as solid tumors by histopathology, and the tumor lesions could be detected or evaluated;
3. Be after standard treatment or who lack effective treatment programs;
4. Patients and their families were willing to participate in the clinical trial and signed the informed consent;
5. Physical status: ECOG score 0-1;
6. Expected survival time > 3 months;
7. HIV antibody negative;Hepatitis b surface antigen negative;Hepatitis c antibody negative;The results of blood routine and coagulation were roughly normal, lymphocyte >0.8×10^9/L, hemoglobin >100g/L, and the pregnancy test of female patients with fertility potential was negative.
8. Left ventricular ejection fraction 50% as indicated by cardiac ultrasound;Upper normal level of serum ALT/AST < 2.5 times;Serum creatinine 1.6mg/dl;Total bilirubin 1.5mg/dl, subject's total bilirubin < 3mg/dl except for Gilberts Syndrome;
9. At least 4 weeks after the last systemic treatment, the patient's toxic and side effects must be restored to grade 1 or lower (except for alopecia or vitiligo).If the subject undergoes minor surgery within 3 weeks prior to enrollment, as long as all toxicity is recovered to level 1 or lower, the subject will meet the enrollment requirements.
10. During the whole study period, patients can regularly visit the enrolled research institutions for relevant detection, evaluation and management;
11. The patient is not allowed to use any anti-tumor drugs or treatments for 4 weeks prior to the infusion of TCR-T cells;
12. Patients' tumor lesions can be obtained by surgery or puncture, and tumor infiltrating T cells can be successfully isolated from the obtained tumor tissue;
13. T cells in patients' peripheral blood can effectively proliferate and expand by at least 10 times in the Pre-culture;
14. The benefits of participating in the clinical trial outweigh the risks,which was evaluated by the researchers base on the status or condition of the patients.

Exclusion Criteria:

1. Any form of primary immunodeficiency disease (such as severe combined immunodeficiency disease);
2. Experiencing moderate to severe infection or possible opportunistic infection;
3. Patients with a history of autoimmunity (e.g., SLE, psoriasis, etc.);
4. Acute systemic infection, coagulation dysfunction or other serious cardiopulmonary diseases;
5. Patients who have is suffering a large amount of glucocorticoid or other immunosuppressive agents within 4 weeks;
6. Be allergic to any drug used in this study;
7. Central nervous system metastases patients with clinically unstable or acute meningitis (except these clinically stable after treatment) Clinical stability needs to be met as follows: 4 weeks at least before the trial treatment, 1) no new brain lesion or no expanded of the original lesions confirmed by MRI); 2) no hormone therapy for at least 2 weeks; 3) neurological symptoms have returned to baseline;
8. Pregnant and lactating women, as well as male and female patients who could not cooperate with contraception during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | At least 45 days
  Keep records the adverse events experienced by subjects in 30 days after the last infusion.

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | one year
  DCR is defined as the proportion of patients with tumor size reduction(CR,PR) and stable (SD) assessed by RECIST 1.1 and iRECIST
overall survival(OS) | two year
  The time from the first injection of Investigational Product until death
progression-free survival(PFS) | two year
  PFS is defined as the time from the first injection of Investigational Product until objective tumor progression or death, whichever occurs first.Assessed by RECIST 1.1 and iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Penghui Zhou, Study Director — Guangzhou FineImmune Biotechnology Co., LTD.
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gaungdong, China

IPD SHARING:
Plan to Share IPD: No